CLINICAL TRIAL: NCT04647071
Title: Study of the Effect of the Consumption of a Combination of Allium Extracts on the Incidence of Symptoms of Respiratory Infections in Healthy Elderly Residents
Brief Title: Allium Extracts on the Incidence of Respiratory Infection Symptoms in Healthy Elderly Volunteers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: DOMCA S.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: C002
Record Dates: First submitted 2020-10-22; First posted 2020-11-30 (Actual); Last update posted 2022-05-23 (Actual); Status verified 2020-11

CONDITIONS: Immunity
Keywords: Garlic; Onion; Immunity
MeSH Terms: interventions — Excipients

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Each volunteer is assigned a "participant number" that will be associated with a pot that will have all the product for the study.
  The "pot number" is the same as the "participant number". The pot does not indicate which product it is carrying.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (Placebo Comparator): Microcrystalline cellulose (9892- Capsules®) up to 400 mg.
  Interventions: Dietary Supplement: Garlic and onion concentrate; Dietary Supplement: Control
- Intervention (Experimental): Garlic concentrated extract plus onion concentrated extract plus microcrystalline cellulose (9892- Capsules®) up to 400 mg.
  Interventions: Dietary Supplement: Garlic and onion concentrate; Dietary Supplement: Control

INTERVENTIONS:
Dietary Supplement: Garlic and onion concentrate — Garlic extract concentrate (equivalent to 2 garlic cloves) and onion extract concentrate (equivalent to 1 onion).
  Other Names: AlioCare
Dietary Supplement: Control — Microcrystalline cellulose
  Other Names: Excipient

SUMMARY:
To analyze the efficacy of daily consumption of a combination of garlic and onion extracts on the incidence of respiratory infection symptoms in healthy elderly volunteers living in a residence.

The duration of symptoms and related medication will also be studied.

DETAILED DESCRIPTION:
It is a controlled, randomized, double-blind, parallel-group nutritional intervention study.

66 healthy elderly volunteers living in a nursing home will be randomly distributed into 2 equal groups: control group and intervention group.

For 36 weeks the volunteers will take the product immediately after lunch. During that time they will maintain their lifestyle and nutritional habits.

Every 4 weeks, the medical team of the residence will review the cases of respiratory diseases of infectious origin of the volunteers.

ELIGIBILITY:
Inclusion Criteria:

* Live in a nursing home with medical services.
* Accept being vaccinated for the flu.
* Freely accepted to participate in the study and sign the informed consent document.
* Have the consent of the family.

Exclusion Criteria:

* Having any disease that affects the development and results of the study.
* Be unable to understand the study and sign voluntarily and freely the informed consent.
* Have a low expectation of compliance with the study protocol.

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 66 (Actual)
Dates: Start 2020-11-16 (Actual); Primary Completion 2021-07-26 (Actual); Study Completion 2022-01-31 (Actual)

PRIMARY OUTCOMES:
Incidence of respiratory symptoms associated with infections. | 36 weeks.
  It will be reviewed if the volunteer has had any symptoms related to respiratory diseases of infectious origin.

SECONDARY OUTCOMES:
Duration of symptoms. | 36 weeks
  If the volunteer has had any symptoms related to respiratory diseases of infectious origin, every 4 weeks duration of these symptoms will be reviewed.
Consumption of medicines. | 36 weeks
  If the volunteer has had any symptoms related to respiratory diseases of infectious origin, every 4 weeks treatment applied will be reviewed.

CONTACTS AND LOCATIONS:
Overall Officials: Carlos Gracián, MD, Principal Investigator — Claret Residence for the Elderly (Granada, Spain).
Locations (1):
- Residencia de Mayores Claret, Granada, Spain